CLINICAL TRIAL: NCT03873662
Title: Biochemical Makers for Outcome Prognostication After Pediatric out-of Hospital Cardiac Arrest: Observational Cohort Trial
Brief Title: Biochemical Makers for Outcome After Pediatric out-of Hospital Cardiac Arrest
Acronym: BIMOPECA
Status: Terminated | Type: Observational
Why Stopped: Low inclusion rate
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: Biomarkers KDAR 2019
Record Dates: First submitted 2019-03-03; First posted 2019-03-13 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Out-Of-Hospital Cardiac Arrest; Pediatric patient; Outcome; Prognostication; Neurologic outcome
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients after out-of hospital cardiac arrest: Pediatric patients after out-of hospital cardiac arrest admitted to Department of pediatric anesthesia and intensive care University hospital in Brno in selected study period with blood sample analysis for neurologic outcome prognostication
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Biochemical markers will be recorded as follows: as soon as possible after the arrival of the patient and insertion of a intravenous line, blood will be drawn for the analysis of arterial blood gases, which are a standard test in patients admitted to emergency department. Blood will be analysed in a bed-side analyzer. Serum lactate and base-excess (BE) will be documented from this blood sample. Another blood sample will be drawn parallelly for biochemical tests which will be sent to the laboratory. These tests standard in patients admitted to emergency department. Serum concentration of NSE and S100B protein will be analysed and recorded from this sample. A sample of blood for the evaluation of the early dynamics of the serum concentration of NSE and S100B will be redrawn after 12 and 48/24 hours after admitting the patient.
  Other Names: Blood biochemical makers analysis

SUMMARY:
This single-center study will validate serum, imaging and clinical markers to determine outcome of pediatric patients early after Out-of-Hospital cardiac arrest (OHCA). Results are expected to add to the field of postresuscitation care of these children. The validation of markers will provide clinicians with the tools to assess the severity of neurological impairment after hypoxic injury to the brain early after OHCA.

DETAILED DESCRIPTION:
Cardiac arrest (CA) is an important cause of mortality and morbidity in pediatric patients. Yearly incidence of CA is 7- 8 cases per 100000 children. Hypoxia is the leading cause of OHCA with up to 1/3 being of respiratory origin, and drowning in ¼ of cases. Up to 2/3 of children admitted to hospitals after OHCA die, with only 16,2% survivors with good neurological outcome. Pediatric cerebral performance category (pCPC) 5, which means persistent coma with patent brainstem reflexes or president vegetative state, or pCPC 6 -brain death is considered a bad outcome in pediatric OHCA survivors.

Early prediction of poor outcome is desirable to avoid futile care and to guide the communication with the relatives of the patient.

There is no published recommendation for the prognostication of outcome of comatose pediatric cardiac arrest survivors. The recommendations for adult patients contains the use of neuron-specific enolase (NSE) and protein S-100B in combination with further predictors in prognosticating the outcome of CA. The remaining problem is to determine a cut-off value, to predict poor outcome (CPC category 5 and 6) with 100% specificity. For this reason, the cut-off values are not included in the recommendations.

Neuron-specific enolase is a glycolytic enzyme localized primarily in the cytoplasma of the neurons. The protein S-100B is a calcium-binding protein specific for the astroglia. Both are sensitive and specific markers for neuronal, respectively astroglial cell death. According to data available in the adult population, serum concentration of NSE and S100B are sensitive and specific markers of traumatic brain injury. High concentration of NSE 3 days after cardiac arrest is a strong predictor of poor outcome. Data regarding the prognostic value of neuronal biomarkers in comatose pediatric CA survivors are scarce.

The aim of the pilot study is to determine the association of the concentration of neuronal biomarkers and the outcome of pediatric CA survivors admitted to the pediatric ICU of the University Hospital Brno. The association will be evaluated individually and in combination with clinical and imaging variables. The basic hypothesis is, that the biochemical, clinical and imaging markers of neurological injury are able to prognosticate poor outcome (pCPC 5-6) with high sensitivity and specificity. The innovation of the study will be the evaluation of the dynamics of serum biomarkers early after CA (first 48 hours).

This is a prospective observational study. All consecutive patients admitted to the ICU of the University Hospital Brno after OHCA and cardiopulmonary resuscitation (CPR), whose parents sign an informed consent will be included. In case the parents will not be present at the time the patient will be admitted, an independent physician will wigh the consent, and the parents consent will be obtained as soon as possible. In case of waiver of consent, the samples will not be included in the final analysis and the patient will be excluded from the study. Patients will be treated according to the actual Guidelines for postresuscitation care. Patients will be treated according to the international guidelines for postresuscitation care. Demographic data will be recorded according to the Utstein Resuscitation Registry Templates for Out-of-Hospital Cardiac Arrest, previously used for the reporting of data on pediatric CA survivors. Clinical parameters, previously shown to be associated with outcomes of patients after OHCA will be recorded. These include: neurological status (level of consciousness as Glasgow coma scale (GCS), reaction of pupils to light, corneal reflex, presence of myoclonus).

Biochemical markers will be recorded as follows: as soon as possible after the arrival of the patient and insertion of a intravenous line, blood will be drawn for the analysis of arterial blood gases, which are a standard test in patients admitted to emergency department. Blood will be analysed in a bed-side analyzer. Serum lactate and base-excess (BE) will be documented from this blood sample. Another blood sample will be drawn parallelly for biochemical tests which will be sent to the laboratory. These tests standard in patients admitted to emergency department. Serum concentration of NSE and S100B protein will be analysed and recorded from this sample. A sample of blood for the evaluation of the early dynamics of the serum concentration of NSE and S100B will be redrawn after 12 and 48/24 hours after admitting the patient.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 weeks -18 years of age
* Child who suffered an out of hospital CA: defined as "Cessation of cardiac mechanical activity as confirmed by the absence of signs of circulation. Includes the following rhythms: pulseless electrical activity (PEA), asystole, ventricular tachycardia, and ventricular fibrillation" with the need od chest compressions.
* Children admitted to the Department of pediatric anesthesia and intensive care
* Children have vascular access for blood draws as part of their standard of care
* Children have a pre-CA Pediatric Cerebral Performance Category (PCPC) score of 1- 3.

Exclusion Criteria:

* Patients with brain injury of other etiologies. (trauma, abscess, tumor, bacterial meningitis)
* Children with do not resuscitate (DNR) status
* Pregnancy
* Metabolic or other disease affecting the brain (eg. refractory epilepsy)

Ages: 14 Days to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pediatric patient after out-of hospital cardiac arrest
Study Population: Pediatric patients after out-of hospital cardiac arrest admitted to Departemnt of pediatric anesthesia and intensive care
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Pediatric cerebral performance category | One year from cardiac arrest
  To evaluate the serum levels of NSE and S100B during first 7 days of hospitalization to determine poor outcome at 1 year post-CA defined as pCPC 5-6
Pediatric cerebral performance category | 3 months from cardiac arrest
  To evaluate the serum levels of NSE and S100B during first 7 days of hospitalization to determine poor outcome at 3 months post-CA defined as pCPC 5-6

SECONDARY OUTCOMES:
Pediatric cerebral performance category | 3 months from cardiac arrest
  To evaluate the association between early dynamics (24 hours from admission) of serum concentration of NSE and S100B in OHCA pediatric patients and Pediatric cerebral performance category scale at 3 months

OTHER OUTCOMES:
Early dynamics of neuronal biomarkers NSE and S100B and association with neurologic outcome | 12 months from cardiac arrest
  To evaluate the association between early dynamics (24 hours from admission) of serum concentration of NSE and S100B in OHCA pediatric patients and Pediatric cerebral performance category scale at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, assoc.Prof.MD.Ph.D, Study Chair — University Hospital Brno
Locations (1):
- University hospital Brno, Brno, State, Czechia

IPD SHARING:
Plan to Share IPD: Undecided